CLINICAL TRIAL: NCT06814379
Title: Rehabilitation of Fatigue in Patients With Post-COVID-19 Syndrome
Acronym: COVIDATE-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Torres Sánchez, PT, PhD, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVIDATE-02
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02

CONDITIONS: Post-COVID-19 Syndrome
Keywords: COVID-19; post-COVID-19 syndrome; fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Fatigue | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Not intervention
- Rehabilitation (Experimental): 30-60 minutes. A total of 3 session/week at home. 4 weeks.
  * Warm-up.
  * Aerobic: walking (20-25 minutes).
  * Strength: (25-30 minutes).
  * Cooling.
  * Education: WHO recommendations.
  Interventions: Behavioral: Rehabilitation
- Virtual reality based rehabilitation (Experimental): 30-60 minutes. A total of 3 session/week (2 sessions at home and 1 session at the University of Granada). 4 weeks.
  The 2 sessions at home will be the same as the sessions in the rehabilitation group (group 2).
  The session at the University of Granada will be done with virtual reality (Nintendo Switch) and will follow the same outline as the rest of the sessions:
  * Warm-up.
  * Aerobic: walking (20-25 minutes).
  * Strength: (25-30 minutes).
  * Cooling.
  * Education: WHO recommendations.
  Interventions: Behavioral: Virtual reality based rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — 30-60 minutes. A total of 3 session/week at home. 4 weeks.
  * Warm-up.
  * Aerobic: walking (20-25 minutes).
  * Strength: (25-30 minutes).
  * Cooling.
  * Education: WHO recommendations.
  Arms: Rehabilitation
Behavioral: Virtual reality based rehabilitation — 30-60 minutes. A total of 3 session/week (2 sessions at home and 1 session at the University of Granada). 4 weeks.
  The 2 sessions at home will be the same as the sessions in the rehabilitation group (group 2).
  The session at the University of Granada will be done with virtual reality (Nintendo Switch) and will follow the same outline as the rest of the sessions:
  * Warm-up.
  * Aerobic: walking (20-25 minutes).
  * Strength: (25-30 minutes).
  * Cooling.
  * Education: WHO recommendations.
  Arms: Virtual reality based rehabilitation

SUMMARY:
More than half of patients with post-COVID-19 syndrome experience fatigue. Rehabilitation is needed to treat this persistent symptom.

The aim of this study is to conduct a rehabilitation intervention to treat patients with post-COVID-19 syndrome who experience persistent fatigue.

DETAILED DESCRIPTION:
* Background: More than half of patients with post-COVID-19 syndrome experience fatigue. Rehabilitation is needed to treat this persistent symptom.
* Objectives: To conduct a rehabilitation intervention to treat patients with post-COVID-19 syndrome who experience persistent fatigue.
* Methodology: Randomized clinical trial. There will be 3 groups.
* Patients will be recruited from the Virgen de las Nieves University Hospital in Granada.
* The evaluation will be carried out at the University of Granada.
* The rehabilitation will be carried out at the University of Granada and/or patient's home.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COVID-19
* post-COVID-19 syndrome
* adults ≥ 18 y < 75 años
* be medically stable
* to be able to walk
* not currently participating in a rehabilitation programme and/or other study.
* fatigue: FSS ≥ 36 puntos
* basic knowledge
* wish to participate in the study and sign the informed consent

Exclusion Criteria:

* patients with severe comorbidities that interfere with the ability to perform the study
* patients with mental, physical or organic problems that under medical criteria may pose a risk to the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Perceived Fatigue | Through study completion, an average of 1 year
  To assess perceived fatigue using the borg modified scale.The scale ranges from 0 to 10, with higher scores indicating greater fatigue perception.
Multidimensional Fatigue | Through study completion, an average of 1 year
  To assess multidimensional fatigue using the multidimensional fatigue inventory MFI-20). The scale comprises five subscales (General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Activity, and Reduced Motivation), each ranging from 4 to 20 points. Higher scores indicate greater fatigue.
Fatigue Severity | Through study completion, an average of 1 year
  To assess fatigue severity using the fatigue severity scale (FSS). The total score ranges from 7 to 63 points, with higher scores indicating greater fatigue severity. A score of ≥36 is considered indicative of significant fatigue.
Fatigue Impact | Through study completion, an average of 1 year
  To assess fatigue impact using the Modified Fatigue Impact Scale (MFIS). Scores range from 0 to 36, with higher scores indicating a greater impact of fatigue on daily activities.

SECONDARY OUTCOMES:
COVID-19 information | Through study completion, an average of 1 year
  To assess information about the date and symptoms when COVID-19 was diagnosed and the COVID-19 Yorkshire Rehabilitation Scale (C19-YRS). The C19-YRS ranges from 0 to 10 per domain (physical, psychological, and functional symptoms). Higher scores indicate greater impairment.
Comorbidities | Through study completion, an average of 1 year
  To assess comorbidities using the Charlson Comorbidity Index (CCI). Scores range from 0 to ≥6, with higher scores indicating greater comorbidity burden.
Dyspnea. The Borg Modified Scale | Through study completion, an average of 1 year
  Ranges from 0 to 10, with higher scores indicating greater dyspnea.
Dyspnea. Dyspnea-12 | Through study completion, an average of 1 year
  Ranges from 0 to 36, with higher scores indicating greater dyspnea severity.
Dyspnea. Modified Medical Research Council (mMRC) Dyspnea Scale | Through study completion, an average of 1 year
  Ranges from 0 to 4, with higher scores indicating greater dyspnea severity.
Pain intensity | Through study completion, an average of 1 year
  To assess pain intensity using the Visual Analogue Scale (VAS). Scores range from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
Psychological status | Through study completion, an average of 1 year
  To assess psychological status using the Hospital Anxiety and Depression Scale (HADS). The scale has two subscales (Anxiety and Depression), each ranging from 0 to 21. Scores of ≥11 on either subscale indicate clinically significant anxiety or depression.
Sleep quality | Through study completion, an average of 1 year
  To assess sleep quality using the Pittsburgh Sleep Quality Index (PSQI). Scores range from 0 to 21, with higher scores indicating poorer sleep quality. A score >5 suggests significant sleep disturbances.
Health-related Quality of life | Through study completion, an average of 1 year
  To assess health-related quality of life using the EuroQol-5D (EQ-5D). Higher scores indicating better quality of life.
Functional status: Post-COVID-19 Functional Status (PCFS) | Through study completion, an average of 1 year
  Ranges from 0 to 4, with higher scores indicating greater functional limitation.
Functional status: Patient-Specific Functional Scale (PSFS) | Through study completion, an average of 1 year
  Scores range from 0 to 10, with higher scores indicating better functional status.
Frailty: Clinical Frailty Scale (CFS) | Through study completion, an average of 1 year
  Ranges from 1 (very fit) to 9 (terminally ill). Higher scores indicate greater frailty.
Frailty: FRAIL Scale | Through study completion, an average of 1 year
  Scores range from 0 to 5, with scores ≥3 indicating frailty.
Physical activity | Through study completion, an average of 1 year
  To assess physical activity using the International Physical Activity Questionnaire (IPAQ). This measure assesses types and intensities of physical activity, yielding results in MET-min/week. Higher values indicate greater physical activity levels.
Exercise capacity: Short Physical Performance Battery (SPPB) | Through study completion, an average of 1 year
  Ranges from 0 to 12, with higher scores indicating better performance.
Exercise capacity: 2-Minute Walk Test | Through study completion, an average of 1 year
  Measures the distance walked in meters; higher values indicate better capacity.
Exercise capacity: One-Legged Stand Test | Through study completion, an average of 1 year
  Measures time in seconds; higher values indicate better balance and strength.
Exercise capacity: Arm Curl Test | Through study completion, an average of 1 year
  Measures the number of arm curls completed in 30 seconds; higher values indicate better upper body strength.
Strength | Through study completion, an average of 1 year
  To assess strength using dynamometry. Results are measured in kilograms (kg), with higher values indicating greater strength.
Motivation for Treatment | Through study completion, an average of 1 year
  15-item Treatment Self-Regulation Questionnaire (TSRQ). Scores range from 1 to 7 per item, with higher scores indicating greater autonomous motivation.
Treatment-Generated Motivation | Through study completion, an average of 1 year
  22-item Intrinsic Motivation Inventory (IMI). Scores range from 1 to 7 per item, with higher scores indicating greater intrinsic motivation.
Satisfaction with the Intervention | Through study completion, an average of 1 year
  5-point Likert scale, with higher scores indicating greater satisfaction.
Overall Perceived Effort | Through study completion, an average of 1 year
  Modified Borg Scale, ranging from 0 to 10, with higher scores indicating greater effort.
Adherence | Through study completion, an average of 1 year
  Monitored via a diary, with adherence reported as the percentage of sessions completed.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Torres Sánchez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No